CLINICAL TRIAL: NCT05778773
Title: OUTcomes Evaluation of Current Therapeutic STrategies for Severe Aortic Valve steNosis anD the agING Population in ITALY
Acronym: OUTSTANDING
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Marco Ranucci, Director of the Cardiovascular Anesthesia and Intensive Care Department, IRCCS Policlinico S. Donato
Other Study IDs: OUSTANDING ITALY
Record Dates: First submitted 2023-03-10; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Aortic Valve Stenosis
Keywords: aortic valve stenosis; aortic valve replacement; transcatheter aortic valve replacement; quality of life; patient registry
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAVR: Patients undergoing aortic valve replacement through the Transcatheter Aortic Valve Replacement procedure.
  For all the patients a set of clinical, anatomical, and procedural details will be obtained and registered. The outcome at the hospital discharge and at the 12-month follow-up will be collected, as well. The quality of life questionnaire will be administered to all the patients at the hospital discharge, at the 12-month follow-up (mandatory), and then at annual base (facultative).
  Interventions: Procedure: TAVR (Transcatheter Aortic Valve Replacement)
- AVR: Patients undergoing aortic valve replacement through conventional open-heart surgery (sternotomy and biological valve implantation).
  For all the patients a set of clinical, anatomical, and procedural details will be obtained and registered. The outcome at the hospital discharge and at the 12-month follow-up will be collected, as well. The quality of life questionnaire will be administered to all the patients at the hospital discharge, at the 12-month follow-up (mandatory), and then at annual base (facultative).
  Interventions: Procedure: AVR (Aortic Valve Replacement)

INTERVENTIONS:
Procedure: TAVR (Transcatheter Aortic Valve Replacement) — Percutaneous aortic valve replacement, also known as percutaneous aortic valve implantation, transcatheter aortic valve implantation or transcatheter aortic valve replacement, is the replacement of the aortic valve of the heart through the blood vessels.
  Other Names: TAVI (Transcatheter Aortic Valve Implantation)
  Groups: TAVR
Procedure: AVR (Aortic Valve Replacement) — Aortic valve replacement is a procedure whereby the failing aortic valve of a patient's heart is replaced with an artificial heart valve through an open-heart surgery.
  Groups: AVR

SUMMARY:
In 2015 the Italian Ministry of Health invited the Cardiac Research Hospitals of Italy to constitute a Cardiac Network. The aim of the network is to facilitate and promote scientific and technological research in the setting of cardiovascular diseases and related risk factors. IRCCS (Scientific Research and Cure Institute) Policlinico San Donato is the responsible hospital for cardiac valve pathologies and has been appointed the leader for the present study.

The non-calcific aortic valve stenosis in the elderly is one of the most frequent cardiovascular diseases. Different therapeutic options are available for treating this condition: medical therapy and follow-up, conventional surgery (including sternotomy and employment of mechanical, biological, or sutureless valves), and transcatheter valve implantation. The uncertainty about the advantages and limitations of the different approaches is still very high.

In this panorama, the concept of mere survival should be replaced by a broader vision of the quality of life. The aim of the present study is to build an Italian registry of aortic valve stenosis in the elderly (age >= 65 years) who, following the current guidelines, would receive a biological aortic valve replacement. The following topics will be evaluated: (i) the results of the different therapeutical options; (ii) the determination of the choice criteria for the different therapeutical options and the verification of the appropriateness, economic and organizational impact for each of them; (iii) the evaluation of the quality of life modifications, periprocedural and at a long follow-up; (iv) the health technology assessment of the applied therapies.

DETAILED DESCRIPTION:
In 2015 the Italian Ministry of Health invited the Cardiac Research Hospitals of Italy to constitute a Cardiac Network. The aim of the network is to facilitate and promote scientific and technological research in the setting of cardiovascular diseases and related risk factors. IRCCS (Scientific Research and Cure Institute) Policlinico San Donato is the responsible hospital for cardiac valve pathologies and has been appointed the leader for the present study.

The proportion of the elderly in the general population is constantly increasing over the last few years and is destined to grow further in industrialized countries, representing a challenge for the sanitary authorities for a number of reasons.

The non-calcific aortic valve stenosis in the elderly is one of the most frequent cardiovascular diseases. Different therapeutic options are available for treating this condition: medical therapy and follow-up, conventional surgery (including sternotomy and employment of mechanical, biological, or sutureless valves), and transcatheter valve implantation (TAVI). The uncertainty about the advantages and limitations of the different approaches is still very high.

In this panorama, mere survival should be replaced by a broader vision of the quality of life. The aim of the present study is to build an Italian registry of aortic valve stenosis in the elderly (age >= 65 years) who, following the current guidelines, would receive a biological aortic valve replacement. The following topics will be evaluated: (i) the results of the different therapeutical options; (ii) the determination of the choice criteria for the different therapeutical options and the verification of the appropriateness, economic and organizational impact for each of them; (iii) the evaluation of the quality of life modifications, periprocedural and at an extended follow-up; (iv) the health technology assessment of the applied therapies.

ELIGIBILITY:
Inclusion Criteria:

* age higher or equal to 65 years;
* aortic valve stenosis that, according to current guidelines, should be treated by a valve replacement;
* written consent to participate.

Exclusion Criteria:

* aortic valve insufficiency not due to stenosis;
* refusal to participate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients hospitalized due to aortic valve stenosis that is to be treated, according to the current guidelines, through a replacement, be it a percutaneous procedure (transcatheter aortic valve replacement) or an open-heart surgery (sternotomy, cardiopulmonary bypass, and biological aortic valve implantation), as agreed between the cardiologist, the surgeon, the anesthesiologist, and the patient.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days after procedure
  Percentage of patients died

SECONDARY OUTCOMES:
Quality of life index | Hospital discharge (average 2 to 7 days after procedure/surgery); 12-month follow-up
  Index of well-being assessed through a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nkomo VT, Gardin JM, Skelton TN, Gottdiener JS, Scott CG, Enriquez-Sarano M. Burden of valvular heart diseases: a population-based study. Lancet. 2006 Sep 16;368(9540):1005-11. doi: 10.1016/S0140-6736(06)69208-8. PMID 16980116
- [Background] Iung B, Vahanian A. Epidemiology of acquired valvular heart disease. Can J Cardiol. 2014 Sep;30(9):962-70. doi: 10.1016/j.cjca.2014.03.022. Epub 2014 Mar 21. PMID 24986049
- [Background] D'Agostino RS, Jacobs JP, Badhwar V, Fernandez FG, Paone G, Wormuth DW, Shahian DM. The Society of Thoracic Surgeons Adult Cardiac Surgery Database: 2019 Update on Outcomes and Quality. Ann Thorac Surg. 2019 Jan;107(1):24-32. doi: 10.1016/j.athoracsur.2018.10.004. Epub 2018 Nov 10. PMID 30423335
- [Background] Mylotte D, Osnabrugge RLJ, Windecker S, Lefevre T, de Jaegere P, Jeger R, Wenaweser P, Maisano F, Moat N, Sondergaard L, Bosmans J, Teles RC, Martucci G, Manoharan G, Garcia E, Van Mieghem NM, Kappetein AP, Serruys PW, Lange R, Piazza N. Transcatheter aortic valve replacement in Europe: adoption trends and factors influencing device utilization. J Am Coll Cardiol. 2013 Jul 16;62(3):210-219. doi: 10.1016/j.jacc.2013.03.074. Epub 2013 May 15. PMID 23684674
- [Background] Cosgrove DM 3rd, Sabik JF. Minimally invasive approach for aortic valve operations. Ann Thorac Surg. 1996 Aug;62(2):596-7. No abstract available. PMID 8694642
- [Background] Cribier A, Eltchaninoff H, Bash A, Borenstein N, Tron C, Bauer F, Derumeaux G, Anselme F, Laborde F, Leon MB. Percutaneous transcatheter implantation of an aortic valve prosthesis for calcific aortic stenosis: first human case description. Circulation. 2002 Dec 10;106(24):3006-8. doi: 10.1161/01.cir.0000047200.36165.b8. PMID 12473543
- [Background] Lababidi Z. Aortic balloon valvuloplasty. Am Heart J. 1983 Oct;106(4 Pt 1):751-2. doi: 10.1016/0002-8703(83)90097-2. No abstract available. PMID 6225323
- [Background] Lababidi Z, Wu JR, Walls JT. Percutaneous balloon aortic valvuloplasty: results in 23 patients. Am J Cardiol. 1984 Jan 1;53(1):194-7. doi: 10.1016/0002-9149(84)90709-4. PMID 6691261
- [Background] Bordoni B, Moretti C, Marrozzini C, Ciuca C, Dall'Ara G, Taffani L, Chiarabelli M, Taglieri N, Berardini A, Guastaroba P, Bacchi-Reggiani ML, Rapezzi C, Marzocchi A, Saia F. Repeated Aortic Balloon Valvuloplasty in Elderly Patients With Aortic Stenosis Who Are Not Candidates for Definitive Treatment. J Invasive Cardiol. 2015 Dec;27(12):E277-84. Epub 2015 Sep 15. PMID 26378413
- [Background] MAGOVERN GJ, CROMIE HW. SUTURELESS PROSTHETIC HEART VALVES. J Thorac Cardiovasc Surg. 1963 Dec;46:726-36. No abstract available. PMID 14099081
- See also: Italian Population Registry — http://www.istat.it/it/files/2014/05/cap4.pdf